CLINICAL TRIAL: NCT01122719
Title: The Best Trial - Brazilian and Italian Evaluation of Safety Using Tacrolimus-eluting Stent With Short-term Dual Antiplatelet Regimen
Brief Title: Brazilian and Italian Evaluation of Safety Using Tacrolimus-eluting Stent With Short-term Dual Antiplatelet Regimen
Acronym: BEST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow inclusion, due to difficulties in obtaining the patients consent for the 2 months invasive follow-up, as required by protocol design.
Sponsor: CID - Carbostent & Implantable Devices (Industry)
Collaborators: Contract research Organization: Cardiovascular Research Center - Sao Paulo, Brazil (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C21002
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Stable Coronary Disease; Unstable Coronary Disease; Documented Silent Ischemia
Keywords: Optima; Tacrolimus; Drug eluting stent
MeSH Terms: interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Drug Eluting Stent

SUMMARY:
To evaluate the safety and efficacy of the Janus OPTIMA Tacrolimus-Eluting Stent (Optima TES, CID) for the treatment of de novo coronary lesions when associated with short-term (two months) dual antiplatelet (aspirin + clopidogrel) regimen.

DETAILED DESCRIPTION:
The present study is a post-market, prospective, international, two-center, single arm study involving 60 patients with single, de novo non-complex coronary lesions.

Enrolled patients will be asked to return for follow-up clinical evaluation at 1, 6, 12 and 24 months. At 3 months there will be an additional follow-up by phone contact.

Furthermore, the first 15 patients should undergo angiographic and OCT follow-up at two months. The remaining 45 patients should undergo angiographic and IVUS follow-up at 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient with >18 years of age;
* Symptoms of stable or unstable angina and/or presence of a positive functional test for ischemia;
* Presence of a single de novo target lesion located in a native coronary vessel suitable for percutaneous treatment with the study stents;
* Acceptable candidate for coronary artery bypass graft(CABG)surgery;
* The subject is willing to sign a written informed consent prior to procedure, and is willing to undergo ALL study protocol follow-ups,including angiographic, IVUS and OCT assessments.
* Single, de novo lesion
* Target lesion located in a major epicardial coronary vessel with reference of 2.5-3.5mm in diameter (by on-line QCA)
* Target lesions ≤19mm in length (by visual estimation) that can be treated (covered) by one single study stent (19 or 24mm in length);
* ≥50% and <100% diameter stenosis;
* TIMI (Thrombolysis In Myocardial Infarction) flow grade ≥2.

Exclusion Criteria:

* Known hypersensitivity or contraindication to tacrolimus, heparin,any required medications including thienopyridines, and contrast media which cannot be adequately pre medicated;
* Patient is a female with childbearing potential;
* Pre-treatment of the target lesion with any devices other than balloon angioplasty;
* Previous brachytherapy in the target vessel;
* Presence of non-target vessel lesions which require staged procedure(s) <30 days of the index procedure;
* Prior CABG surgery to target vessel;
* Previous percutaneous coronary intervention (PCI) or CABG surgery <30 days to the index procedure date;
* Acute myocardial infarction <3 days, with cardiac enzyme elevation including total creatine kinase (CK) >2 times the upper normal limit value and/or CK-MB above the upper normal limit value within the past 72 hours;
* CK and/or CK-MB levels elevated above the upper normal limit value at the time of the index procedure;
* Documented left ventricular ejection fraction <30%;
* Renal insufficiency determined by a baseline serum creatinine >2.0 mg/dl;
* Thrombocytopenia with a baseline platelet count <100,000 cells/mm3;
* Anemia with baseline hemoglobin <10g/dL;
* Extensive peripheral vascular disease or extreme anticoagulation that precludes safe >5 French sheath insertion;
* History of bleeding diathesis, coagulopathy, or refusal of blood transfusions;
* Patients has suffered a stroke, transient ischemic attack (TIA),or cerebrovascular accident (CVA) within the past 6 months;
* Significant gastrointestinal or genitourinary bleed within the past 6 months;
* Patient is a recipient of a heart transplant;
* Any elective surgical procedure is planned within 12 months of the index procedure;
* Known illness or any serious clinical condition with life expectancy <2 years;
* Participation in the active or follow-up phase of any other clinicaltrial within 6 months;
* Impossibility to comply with anti-platelet therapy during the study clinical follow-up;
* Any impossibility to comply with all protocol follow-ups.
* Target lesion or vessel with angiographic evidence of moderate or severe calcification;
* Presence of severe tortuosity;
* Presence of severe angulation (>60o);
* Presence of intraluminal thrombus;
* Target lesion involving a bifurcation (side branch ≥2.0mm);
* Target lesion located in the left main stem;
* Aorto-ostial lesion location;
* Target lesion involving a side branch with reference diameter≥2.0mm;
* Presence of a significant stenosis (>40%) in the target vessel either proximal or distal to the target lesion that will be untreated;
* Previous placement of a stent within 10mm of the target lesion;
* Total occlusion (TIMI flow grade 0 or 1);
* Target lesion located in an arterial or vein graft;
* Target lesion due to in-stent restenosis;
* Coronary anatomy unsuitable for percutaneous treatment with implantation of the available study stents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
In-stent late lumen loss | 8-month

SECONDARY OUTCOMES:
All-cause and cardiac mortality; | up to 24 months
Myocardial infarction (MI): Q-wave and non-Q-wave, cumulative and individual | up to 24 months
Major Adverse Cardiac Event (MACE) defined as a composite of cardiac death, MI (Q wave or non-Q wave), emergent coronary artery bypass surgery (CABG), or target lesion revascularization (TLR) by repeat PTCA or CABG | up to 24 months
Rate of stent thrombosis using ARC definition of definite and probable stent thrombosis and categorized as early, late or very late | up to 24 months
Stent strut coverage assessed by OCT | 2 months
Late acquired incomplete stent apposition by IVUS | 8-month
In stent & In segment angiographic parameters | 8-month
Clinically Driven TLR | up to 24 months
Clinically Driven TVR | up to 24 months
Target Lesion Failure (TLF) defined as cardiac death, MI and ischemic Target Lesion Revascularization (TLR) | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Marco Valgimigli, Dr, Principal Investigator — Azienda Ospedaliero Universitaria di Ferrara - Italy; Alexandre Abizaid, Dr, Principal Investigator — Instituto Dante Pazzanese de Cardiologia
Locations (2):
- Istituto Dante Pazzanesw, São Paulo, Brazil
- Azienda Ospedaliera Universitaria di Ferrara, Ferrara, Italy